CLINICAL TRIAL: NCT06390332
Title: Inclusive Practices for Gender Minority College Students to Reduce Sexual Violence and Heavy Drinking
Brief Title: Centering Gender Affirming Resources in Higher Education
Acronym: CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Opportunity Fund (Unknown)
Responsible Party: Principal Investigator, Elizabeth Miller, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22040105; R01AA023260-07W1 (NIH)
Record Dates: First submitted 2024-04-17; First posted 2024-04-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sexual Violence; Drinking Heavy
Keywords: Transgender; Gender Minorities
MeSH Terms: interventions — Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giving Information for Trauma Support and Safety (GIFTSS) Training (Active Comparator): Training for college health center clinicians and staff in implementation of GIFTSS
  Interventions: Behavioral: Giving Information for Trauma Support and Safety (GIFTSS) Training
- GIFTSS Training and Centering gender Affirming Resources in higher Education (CARE) Learning Modules (Experimental): Training for college health center clinicians and staff in implementation of GIFTSS combined with CARE's trans learning modules to support implementation with gender diverse service users.
  Interventions: Behavioral: Giving Information for Trauma Support and Safety (GIFTSS) Training; Behavioral: Centering gender Affirming Resources in higher Education (CARE) Learning Modules

INTERVENTIONS:
Behavioral: Giving Information for Trauma Support and Safety (GIFTSS) Training — Training for college health center staff and clinicians on GIFTSS intervention which is a universal education and brief counseling to address sexual violence prevention and intervention.
Behavioral: Centering gender Affirming Resources in higher Education (CARE) Learning Modules — Training for college health center clinicians and staff on trans and gender diverse (TGD) affirming clinical practices in addition to sexual violence and alcohol abuse prevention that is inclusive of TGD service users
  Arms: GIFTSS Training and Centering gender Affirming Resources in higher Education (CARE) Learning Modules

SUMMARY:
Centering gender Affirming Resources in higher Education (CARE) project is nested within the parent study "Reducing Alcohol Involved Sexual violence in higher Education" (RAISE; R01 AA023260; NCT05185440). CARE is a pilot cluster-randomized trial that centers trans and gender diverse (TGD) students who are at elevated risk for SV and hazardous drinking. CARE tests a novel college health and counseling center (CHC) training program designed to improve provider knowledge about TGD individuals, increase their self-efficacy and use of trans-inclusive practices. This includes an evaluation of the feasibility, acceptability, appropriateness, and usability of CARE's training intervention for college health and counseling center providers. This research will produce the first rigorously evaluated TGD-focused CHC provider training which has the potential to increase the accessibility of CHC's for TGD university students- ultimately lowering rates of alcohol use and SV among this disproportionately impacted population.

DETAILED DESCRIPTION:
"Centering gender Affirming Resources in higher Education (CARE)" expands upon RAISE's (R01 AA023260) cluster-randomized controlled trial across 28+ college campuses that is evaluating harm reduction interventions to reduce risk for sexual violence (SV) among undergraduate college students receiving care from college health and counseling centers (CHCs). A previous study by this research team found that students identifying as transgender or gender diverse (TGD) report particularly high lifetime prevalence of SV that is associated with greater odds of binge drinking compared to students not exposed to SV. Compounding these vulnerabilities, TGD students face high rates of discrimination on university campuses that drive heavy alcohol use and SV inequities, and lead to distrust of potential support resources like CHCs. CARE enhances RAISE's intervention by employing community-partnered methodologies to develop a training for CHC providers designed specifically to increase their competence in addressing TGD students' health needs with a focus on alcohol use and SV. The training involves a brief e-learning (asynchronous) intervention aimed at improving providers' knowledge and attitudes about TGD individuals, skills in delivering competent and affirming care, and knowledge of and self-efficacy to use TGD-inclusive practices. This trial will assess the feasibility, acceptability, appropriateness, and usability of CARE's training intervention in 15 randomized CHC sites from the parent study (Aim 1). The study will examine CHC provider knowledge and attitudes about TGD individuals, and their knowledge, self-efficacy, and use of TGD-inclusive practices with follow-up at 4-6 months (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Those who are seeing undergraduate students at health and counseling appointments as a provider.
* Providers may include counselors, clinicians, nurses, health educators, medical assistants, social workers, advocates, and administrators.

Exclusion Criteria:

* A college health or counseling center provider that does not interface with students.
* A college health or counseling center provider not participating in the RAISE study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Provider perception of intervention feasibility | Immediately after CARE training completion
  Domain: Provider-Perceived Feasibility Specific Measurement: Feasibility of Intervention Measure (FIM). Specific Metric: End value Method of Aggregation: Mean score, range 1-5 cutoff mean score > 4, higher score indicates greater feasibility
Provider perception of intervention acceptability | Immediately after CARE training completion
  Domain: Provider-Perceived Acceptability Specific Measurement: Acceptability of Intervention Measure (AIM) Specific Metric: End value Method of Aggregation: Mean score, range 1-5, cutoff mean score > 4, higher score indicates greater acceptability
Provider perception of intervention appropriateness | Immediately after CARE training completion
  Domain: Provider-Perceived Appropriateness Specific Measurement: Intervention Appropriateness Measure (IAM) Specific Metric: End value Method of Aggregation: Mean score, range 1-5 , cutoff mean score > 4, higher score indicates greater appropriateness
Provider perception of intervention usability | Immediately after CARE training completion
  Domain: Provider-Perceived Usability Specific Measurement: System Usability Scale (SUS) Specific Metric: End value Method of Aggregation: Mean score, range 1-5 , cutoff mean score > 4, higher score indicates greater usability

SECONDARY OUTCOMES:
Knowledge and attitudes about TGD individuals. | Baseline- Before taking CARE training
  Domain: Assessing provider knowledge, attitudes, and beliefs about transgender people Specific Measurement: Transgender Knowledge, Attitudes, and Beliefs (T-KAB) scale Specific Metric: End value Method of Aggregation: Mean score, range 1 to 4, 4 indicating favorable attitudes and beliefs towards transgender people
Knowledge and attitudes about TGD individuals. | At 6 months
  Domain: Assessing provider knowledge, attitudes, and beliefs about transgender people Specific Measurement: Transgender Knowledge, Attitudes, and Beliefs (T-KAB) scale Specific Metric: Change from baseline Method of Aggregation: Mean score, range 1 to 4, 4 indicating favorable attitudes and beliefs towards transgender people
Attitudes concerning transphobia | Baseline- Before taking CARE training
  Domain: Assessing provider's attitudes regarding transphobia Specific Measurement: Transphobia Scale Specific Metric: End value Method of Aggregation: Mean score, range 1 to 7, 7 indicating a lesser degree of transphobia
Attitudes concerning transphobia | At 6 months
  Domain: Assessing provider's attitudes regarding transphobia Specific Measurement: Transphobia Scale Specific Metric: Change from baseline Method of Aggregation: Mean score, range 1 to 7, 7 indicating a lesser degree of transphobia
Human value of transgender people | Baseline- Before taking CARE training
  Domain: Assessing how providers view the human value of transgender people Specific Measurement: Transgender Attitudes and Beliefs Scale (TABS) Specific Metric: End value Method of Aggregation: Mean score, range 1 to 7, 7 indicating trans and gender diverse people hold high human value
Human value of transgender people | At 6 months
  Domain: Assessing how providers view the human value of transgender people Specific Measurement: Transgender Attitudes and Beliefs Scale (TABS) Specific Metric: Change from Baseline Method of Aggregation: Mean score, range 1 to 7, 7 indicating trans and gender diverse people hold high human value
Use of TGD-inclusive practices | Baseline- Before taking CARE training
  Domain: Use of transgender and gender diverse-inclusive practices Specific Measurement: The Lesbian, Gay, Bisexual, and Transgender Development of Clinical Skills Scale (LGBT-DOCSS) Specific Metric: End value Method of Aggregation: Mean score, range 1 to 7, 7 indicating high preparedness and knowledge to work with transgender patients
Use of TGD-inclusive practices | At 6 months
  Domain: Use of transgender and gender diverse-inclusive practices Specific Measurement: The Lesbian, Gay, Bisexual, and Transgender Development of Clinical Skills Scale (LGBT-DOCSS) Specific Metric: Change from baseline Method of Aggregation: Mean score, range 1 to 7, 7 indicating high preparedness and knowledge to work with transgender patients
Trans-Inclusivity in professional settings | Baseline- Before taking CARE training
  Domain: Assessing how trans-inclusive providers are in their practice Specific Measurement: The Trans-Inclusive Provider Scale (TIPS) Specific Metric: End value Method of Aggregation: Mean score, range 1 to 5, 5 indicating high trans-inclusivity in care practices)
Trans-Inclusivity in professional settings | At 6 months
  Domain: Assessing how trans-inclusive providers are in their practice Specific Measurement: The Trans-Inclusive Provider Scale (TIPS) Specific Metric: Change from Baseline Method of Aggregation: Mean score, range 1 to 5, 5 indicating high trans-inclusivity in care practices
Social desirability | Baseline- Before taking CARE training
  Domain: Measure of social desirability Specific Measurement: Marlowe- Crowne Social Desirability Scale Specific Metric: End Value Method of Aggregation: True and false questions, summary score from 0 to 1
Social desirability | At 6 months
  Domain: Measure of social desirability Specific Measurement: Marlowe- Crowne Social Desirability Scale Specific Metric: Change from Baseline Method of Aggregation: True and false questions, summary score from 0 to 1
Self-Efficacy to use trans and gender affirming practices | Baseline- Before taking CARE training
  Domain: Self-efficacy to use trans and gender affirming practices Specific Measurement: Investigator Developed Specific Metric: End value Method of Aggregation: Mean score, range 1 to 5, 5 indicating greater self-efficacy to use trans-affirming practices
Self-Efficacy to use trans and gender affirming practices | At 6 months
  Domain: Self-efficacy to use trans and gender affirming practices Specific Measurement: Investigator Developed Specific Metric: Change from baseline Method of Aggregation: Mean score, range 1 to 5, 5 indicating greater self-efficacy to use trans-affirming practices

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, PhD, Principal Investigator — Principal Investigator
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after end of study
Access Criteria: data uploaded to NDA
URL: http://nda.nih.gov/